CLINICAL TRIAL: NCT03719716
Title: Early Support in Primary Care for People Starting Treatment for Cancer
Acronym: GI-ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: NHS Fife (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AC18066
Record Dates: First submitted 2018-09-17; First posted 2018-10-25 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Pancreas; Cancer of Stomach; Cancer of Esophagus
Keywords: Oncology; Palliative Care; Primary care; Care planning
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomised automatically by the local trials unit and allocated a study number. This will be used in all statistical analyses and other quantitative data analysis including the questionnaires. The study researcher will know the identity of the participants she interviews and the qualitative analysis cannot be blinded although all data generated will be anonymised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early support group (Experimental): This group receive the Anticipatory care planning letter to take to their GP and the GP receives a copy of the Scottish Anticipatory Care Planning information leaflet and a short communication guide about ACP.
  Interventions: Other: Anticipatory care planning letter
- Usual care group (No Intervention): No change to standard care from oncology services and primary care

INTERVENTIONS:
Other: Anticipatory care planning letter — Patient letter to take to GP and GP literature
  Arms: Early support group

SUMMARY:
This is a feasibility, randomised controlled trial (RCT) of a person-centred care planning intervention involving patients recently diagnosed with a poor prognosis cancer who are starting a palliative oncology treatment in a Scottish regional cancer centre.

DETAILED DESCRIPTION:
This study will evaluate the feasibility and acceptability of an early 'palliative care' intervention consisting of anticipatory care planning coordinated in primary care that is systematically triggered when patients with poor prognosis gastrointestinal cancers start palliative oncology treatment.

Patients will be identified and invited to participate during their assessment and treatment planning by the cancer care clinicians. A screening log will record eligible cases. Patients who consent will be randomised to receive a letter about the benefits of early anticipatory care planning to take to their preferred general practitioner to help trigger earlier support by their primary care team. Control patients receive usual care. All study patients will be asked to complete 3 questionnaires (EuroQol EQ-5D-5L (full title of tool), ICECAP Supportive Care Measure (full title of tool), and CollaboRATE (full title of tool) for shared decision-making) at baseline, 6, 12, 24 and 48 weeks. A purposive sub-sample of patients, family carer and general practitioner (GP) triads will be invited for interview at around 6 and 20 weeks to explore their experiences of trial participation, their illness and care. Health service use will be recorded including hospital admissions, oncology treatment, palliative care referral, time and place of death or survivorship.

ELIGIBILITY:
Inclusion Criteria:

* People with advanced, inoperable oesophageal, gastric or pancreatic cancers
* People being offered palliative chemotherapy and/or radiotherapy

Exclusion Criteria:

* People too ill to participate or give informed consent.
* Patient who are not fit for oncology treatment or who opt for best supportive care.
* People with other life-limiting conditions likely to cause death within 6 months.
* People with moderate to severe cognitive impairment that precludes completions of questionnaires or participation in interviews.
* People unable to give informed consent or communicate by telephone with the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life: EuroQol EQ-5D-5L | Baseline to 48 weeks or death
  Health related quality of life assessed using the EuroQol EQ-5D-5L.
  The EQ-5D-5L has 2 components:
  There is a descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The EQ VAS (visual analogue scale) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
  The users guide gives details of the scoring system: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L_UserGuide_2015.pdf

SECONDARY OUTCOMES:
Trial feasibility assessment: conversion rate | Baseline to 48 weeks or death for last recruited participant
  Screening to consent conversion rate

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Boyd, PhD, Principal Investigator — The University of Edinburgh/ NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, NHS Lothian, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All non-person identifiable data will be collected and stored to allow it to be archived and shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Up to 10 years post study
Access Criteria: During study data will not be shared just the supporting information. After study storage will be arranged by The University of Edinburgh